CLINICAL TRIAL: NCT06189729
Title: Facilitating Routine HIV Testing Among MSM by a Subscription-based HIV Self-test Distribution Model: a Stepped Wedge Randomised Controlled Trial
Brief Title: Facilitating Routine HIV Testing Among MSM by a Subscription-based Self-test Distribution Model
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz Ho Kwan, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 22-0406
Record Dates: First submitted 2023-11-21; First posted 2024-01-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hiv
Keywords: men who have sex with men; hiv self-test
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge trial. In this study, the 1-year observation period is divided into four three-month intervals. All sequences would start with a control period. The three sequences would cross over to the intervention at Month 3, 6, and 9, respectively. All participants would therefore eventually receive intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cluster 1 (Other): Participants will receive text reminders at Month 0 only. They will receive an HIV self-test at Months 3, 6, 9 and 12, upon submission of the self-test result.
  Interventions: Behavioral: Text reminder; Behavioral: HIV self-test
- Cluster 2 (Other): Participants will receive text reminders at Months 0 and 3. They will receive an HIV self-test at Months 6, 9 and 12, upon submission of the self-test result.
  Interventions: Behavioral: Text reminder; Behavioral: HIV self-test
- Cluster 3 (Other): Participants will receive text reminders at Months 0, 3 and 6. They will receive an HIV self-test at Months 9 and 12, upon submission of the self-test result.
  Interventions: Behavioral: Text reminder; Behavioral: HIV self-test

INTERVENTIONS:
Behavioral: Text reminder — Participants will receive trimonthly text reminders through instant messaging mobile applications or short message service.
Behavioral: HIV self-test — Participants will receive trimonthly text messages asking them to choose a pickup point run by the delivery company to collect the free HIV self-test. Upon receiving the delivery instruction, the self-test kit with bilingual (Chinese and English) instructions would be delivered to the designated location.

SUMMARY:
The goal of this stepped wedge trial is to assess if a subscription-based HIV self-test distribution model could facilitate routine HIV testing in the men who have sex with men community. The main questions it aims to answer are the effectiveness of the model in enhancing routine HIV testing and its acceptability in the community. The 1-year observation period would be divided into control and intervention period. Participants will be reminded to get HIV tested via instant messaging apps or short message service during the control period. During the intervention period, the researchers will deliver an HIV self-test to the participants. Researchers will compare the testing rate between the two periods to see if the intervention can facilitate HIV testing.

DETAILED DESCRIPTION:
Participants would be assigned randomly to a sequence group and crossed over from the control to intervention. In this study, the 1-year observation period is divided into four three-month intervals. All sequences would start with a control period. The three sequences would cross over to the intervention at Month 3, 6, and 9, respectively. All participants would therefore eventually receive intervention. The investigators adopt an mHealth approach for both control and intervention. Based on the results of a previous study that text messages through short message service (SMS) and instant messing (IM) apps are acceptable and feasible in promoting HIV self-management, participants during the control period would receive trimonthly text reminders through their designated IM app or SMS. The message would invite them to get HIV tested with free VCT service provider information. After 14 days, a follow-up message with the link to an online survey would be sent to enquire whether the participants had been tested or not. Participants during the intervention period would receive a trimonthly text messages asking them to choose a pickup point run by the delivery company to collect the free HIVST. Upon receiving the delivery instruction, the HIVST with bilingual (Chinese and English) instructions would be delivered to the designated location. Participants would be asked to perform the self-test and return the photographed result within 14 days. Similarly, after 14 days, a follow-up message with the link to an online survey would be sent to ask them to upload the photo of the test result. The uploaded images would be verified by the research team who are experienced in reading HIVST results both online and offline. Follow-up confirmation testing and medical service referral would be offered if the result was indeterminate or suspected to be positive. If the results were not returned after 14 days, an exit survey would be sent to the participants through IM apps or SMS.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18 years or above
* be biologically male
* have ever had sex with another men
* have more than 1 male sex partners in the past 6 months
* normally reside in Hong Kong
* be able to communicate in written and spoken Chinese or English

Exclusion Criteria:

* previously HIV diagnosis
* unable or unwilling to give informed consent, to complete the questionnaires, to receive text messages as scheduled and when necessary, and to provide the mobile phone number to receive text messages for reminders and delivery notices

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of HIV tests performed with result returned | Month 3 to Month 12
  Number of HIV self-test results returned divided by the total number of HIV self-tests delivered
Retention rate | Month 12
  Proportion of participants completed the questionnaire at Month 12

SECONDARY OUTCOMES:
HIV incidence | Month 3 to Month 12
  Dividing the number of laboratory confirmed HIV-positive results by the total number of person-years
Linkage to care rate | Month 3 to Month 12
  The proportion of tests requiring further confirmation and medical service referral.
Single ease question | Month 3 to Month 12
  In a scale of 1-7, how easy or difficult was the task was?
Net promoter score | Month 3 to Month 12
  In a scale of 0-10, how likely would the participant recommend this model to their peers?
System usability scale | Month 3 to Month 12
  There are ten 5-point Likert scale questions. The scores would be summed and multiply by a factor of 2.5 according to the formula to come up with the score between 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Ho Kwan, PhD, Principal Investigator — Jockey Club School of Public Health and Primary Care
Locations (1):
- Stanley Ho Centre for Emerging Infectious Diseases, Shatin, Hong Kong